CLINICAL TRIAL: NCT03781141
Title: Absorbable Versus Non-Absorbable Suture in Carpal Tunnel and Trigger Finger Wound Closure
Brief Title: Wound Closure Study in Carpal Tunnel and Trigger Finger Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Peter C. Rhee, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 18-004267
Record Dates: First submitted 2018-11-14; First posted 2018-12-19 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Carpal Tunnel Syndrome; Trigger Finger
MeSH Terms: conditions — Carpal Tunnel Syndrome; Trigger Finger Disorder

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Blinded assessment for wound healing
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Absorbable suture (Experimental): Wound closure with absorbable suture.
  Interventions: Procedure: Wound closure
- Non-absorbable suture (Active Comparator): Wound closure with non-absorbable suture.
  Interventions: Procedure: Wound closure

INTERVENTIONS:
Procedure: Wound closure — Comparison of two wound closures

SUMMARY:
Does a difference in patient satisfaction and cosmetic outcome exist between wound closure with absorbable or non-absorbable sutures.

DETAILED DESCRIPTION:
The study will involve randomizing patients to wound closure with absorbable or non-absorbable sutures. We will if scar formation (symptoms and aesthetics) if different between the two types of closures as determined by the patient and observer scar assessment scale version 2.0 (POSAS) and the patient-rated wrist/hand evaluation (PRWHE), between absorbable and non-absorbable suture for wound closure of open carpal tunnel release and trigger finger pulley release.

ELIGIBILITY:
Inclusion Criteria:

* Any patient greater than or equal to 18 years of age.
* Any patient undergoing primary open carpal tunnel release or primary trigger finger pulley release

Exclusion Criteria:

* Any patient identified outside of the proposed study time period.
* Any patient receiving revision surgery
* Patients who have had prior ipsilateral palmar or finger surgery
* Patients with Dupuytren's disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2019-12-01 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Scar formation with the Patient and Observer Scare Assessment Scale | 1 year
  Blinded scar assessment utilizing the patient and observer scar assessment scale version 2.0 (POSAS).
  The POSAS is scored from the perspective of the patient and a blinded observer independently. Scores range from 1 to 10 with 1 indicating normal skin and 10 indicating the worst scar imaginable. The 1 to 10 scoring is performed in 6 domains of various scar characteristics to obtain a total score ranging from 10 to 60. Additionally, there is an overall scar appearance score that ranges from 1 to 10 with 1 indicating normal skin and 10 indicating the worst scar imaginable.

CONTACTS AND LOCATIONS:
Overall Officials: Peter C Rhee, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials